CLINICAL TRIAL: NCT07306143
Title: Prediction of Pressure Injury Risk in the Intensive Care Unit: A Comparative Analysis of Data Mining Algorithms in a Single-Center Retrospective Cohort
Brief Title: Prediction of Pressure Injury Risk in ICU Using Data Mining
Acronym: ICU
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-SBF-NSY-2025
Record Dates: First submitted 2025-12-07; First posted 2025-12-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pressure Injury
Keywords: Pressure injury risk; Data mining; Machine learning; Retrospective study; Risk prediction
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patient Cohort: Adult patients who will be hospitalized in the intensive care unit between October 10, 2020 and October 10, 2025. No interventions will be applied, and all data will be obtained from existing medical records.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a retrospective observational study. No interventions will be applied. All data will be obtained from existing medical records.

SUMMARY:
This study is a retrospective record review conducted among adult patients hospitalized in the intensive care unit of a tertiary hospital between October 10, 2020, and October 10, 2025. The aim of the study is to predict the risk of pressure injury development using demographic, clinical, laboratory, and nursing care-related variables by applying multiple data mining algorithms. No intervention, treatment, or patient contact will occur. All data will be extracted from existing electronic and paper-based medical records and will be fully anonymized prior to analysis. The study poses no risk to participants and will be conducted with approval from the institutional review board or ethics committee.

DETAILED DESCRIPTION:
This observational study uses a retrospective cohort design to analyze the clinical, demographic, laboratory, and nursing documentation records of adult intensive care unit (ICU) patients hospitalized between October 10, 2020, and October 10, 2025. The purpose of the study is to identify factors associated with the development of pressure injury and to compare the predictive performance of multiple data mining and machine learning algorithms, including logistic regression, decision trees, random forest, support vector machines, and gradient boosting models.

Data collection will involve reviewing archived ICU records, patient files, and nursing observation forms. No new data will be collected directly from patients, and no medical interventions or prospective follow-up will be performed. All extracted data will be fully anonymized prior to analysis. The study will be conducted in accordance with ethical principles and has been approved by the Bolu Abant Izzet Baysal University Non-Interventional Clinical Research Ethics Committee.

The expected outcome of this study is to identify the most accurate predictive model for pressure injury risk and to support clinical decision-making processes by contributing to early prevention strategies in the ICU.

ELIGIBILITY:
Inclusion Criteria

* Patients hospitalized in the intensive care unit between October 10, 2020, and * October 10, 2025
* Adult patients aged 18 years and older
* Length of intensive care unit stay of at least 24 hours
* Availability of complete and accessible electronic or paper-based medical records

Exclusion Criteria

* Patients younger than 18 years
* Intensive care unit stay shorter than 24 hours Incomplete, missing, or inconsistent electronic or paper-based medical records
* Presence of a pressure injury diagnosed before or at the time of intensive care unit admission
* Inability to extract pressure injury-related data from medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older who were hospitalized in the intensive care unit (ICU) of a tertiary public hospital between October 10, 2020, and October 10, 2025 will be included in this retrospective observational study. The study population includes patients with a minimum ICU stay of 24 hours and complete, accessible electronic or paper-based medical records. Patients with missing or inconsistent medical record data or with a pressure injury diagnosed before or at the time of ICU admission will be excluded. All data will be collected retrospectively from existing medical records.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Prediction accuracy of pressure injury development | 10 October 2020 to 10 October 2025
  The primary outcome is the predictive accuracy of data mining algorithms in identifying the risk of developing pressure injury among patients hospitalized in the intensive care unit (ICU). Accuracy metrics such as the area under the receiver operating characteristic curve (AUC), sensitivity, specificity, precision, recall, and F1-score will be calculated using retrospective medical record data.

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Can Çiçek, Assoc. Prof., PhD, Principal Investigator — Abant Izzet Baysal University
Locations (2):
- Turkey (Türkiye) (2):
  - Bolu Izzet Baysal State Hospital, Bolu, Bolu
  - Bolu Izzet Baysal State Hospital, Merkez, Bolu

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study uses retrospective clinical records that contain sensitive personal health information. In accordance with institutional policies, ethical committee approval, and national data protection regulations (KVKK), IPD cannot be made publicly available. Only aggregated and de-identified results will be provided in publications.